CLINICAL TRIAL: NCT06685419
Title: Effects of Natural Propolis Extract-Containing Chewing Gum on Dental Plaque Accumulation and Gingivitis
Brief Title: Propolis Containing Chewing Gum and Gingivitis
Status: Completed | Type: Observational
Sponsor: naksaka (Other)
Responsible Party: Sponsor-Investigator, naksaka, Assistant Professor, Istanbul Medipol University Hospital
Organization: Istanbul Medipol University Hospital (Other)
Other Study IDs: IstanbulMUH1
Record Dates: First submitted 2024-11-11; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Gingivitis
Keywords: Propolis; Gingivitis; Oral health
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Group: Placebo gum will be used to reduce plaque index scores 5 times a day, after and between meals, for a total of 3 weeks.
- Test Group/Propolis-containing gum group: Propolis-containing gum will be used to reduce plaque index scores 5 times a day, after and between meals, for a total of 3 weeks.
  Interventions: Other: Propolis containing gum

INTERVENTIONS:
Other: Propolis containing gum — Patients with moderate gingivitis will be asked to use gum containing propolis 5 times a day for a total of 3 weeks.
  Groups: Test Group/Propolis-containing gum group

SUMMARY:
Propolis is a natural, non-toxic, sticky substance produced by honeybees that can kill bacteria, fungi, and larvae invading the beehive. It has been used in the treatment of infections and healing of wounds and burns for years. This study evaluated the effects of chewing gum containing pure propolis on plaque accumulation and gum disease in patients who brushed their teeth regularly.

DETAILED DESCRIPTION:
Plaque is the primary etiological factor of periodontal diseases and as a result, inflammation of the gingiva can clinically lead to irreversible consequences such as bone and attachment loss and even tooth loss. Removing the plaque is the most important criterion in preventing inflammation. Plaque should be removed by brushing and the use of interface cleansing agents such as dental floss. However, it has been reported in studies that manually brushing teeth reduces plaque by 70%.

Propolis, which has anti-inflammatory effects, has been used for years in the treatment of infections and wound healing. Propolis has been used and studied in dental applications such as reduction of dentin sensitivity, prevention of dental caries, treatment of oral mucositis caused by chemotherapy, treatment of gingival diseases and replantation of avulsed teeth. Therefore, we hypothesized that daily pure propolis containing chewing gum can improve periodontal results in gingivitis patients by reducing plaque accumulation. The purpose of this double-blind, randomized, placebo-controlled trial was to evaluate the effectiveness of chewing gum containing pure propolis in addition to mechanical treatment.

This study was planned as a double-blind, parallel design, randomized-placebo-controlled study. The sample size was calculated minimum 24 with 80% power. Considering the possible drop-outs, our study will consist of two groups (test and placebo), each of which includes 30 participants. The test group will chew the gum containing propolis 5 times a day for 10 minutes. Participants in the placebo group will chew the placebo gum, prepared with the same color, appearance and consistency, 5 times a day for 10 minutes. Both groups will be asked to chew the gums for 3 weeks after meals (3 main meals - 2 snacks)

Baseline periodontal records including plaque index and gingival index of all participants will be taken and scaling and root planing will be performed. All periodontal treatments and measurements will be made by a single periodontologist. Periodontal measurements will be performed on 4 surfaces of all teeth (mesio-buccal, mid-buccal, disto-buccal, mid-lingual) using a Williams periodontal probe. Patients who are eligible to participate in the study will be assigned to the placebo or test group by the closed envelope method.

Plaque index, gingival index, temporomandibular joint pain, sensation change, taste change will be evaluated using the Visual Analogue Scale (VAS). All parameters will be evaluated 1 week, 2 weeks and 3 weeks after the procedure. The data recorded in the form will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy
* Has at least 20 teeth in his/her mouth.

Exclusion Criteria:

* Smokers
* ongoing orthodontic treatment
* Allergy to the honey and honey-bee products
* periodontal therapy in the last 6 months.
* Pregnancy and breastfeeding
* Use of antibiotics or another drugs in the last three months,
* Presence of subgingival caries or infection that will affect brushing
* Patients who were not willing to participate in the study

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants will be selected from the patients who apply to Istanbul Medipol University for gingival treatment.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-04-06 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
Plaque index | 1 month
  Change in plaque index
Gingival index | 1 month
  Change in plaque index

SECONDARY OUTCOMES:
Temporomandibular joint pain | 1 month
  Temporomandibular joint pain
Changes in taste | 1 month
  Changes in taste

CONTACTS AND LOCATIONS:
Overall Officials: Nurcan Altas, Principal Investigator — Istanbul Medipol Univeristy
Locations (1):
- Istanbul Medipol University, Istanbul, Esenler, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No